CLINICAL TRIAL: NCT04678414
Title: Infertility Survey Among Reproductive Age Women With Gynecological and Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0477; NCI-2020-08295 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0477 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Endometrial Carcinoma; Female Reproductive System Disorder; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Stage I Uterine Corpus Cancer AJCC v8; Stage IA Cervical Cancer AJCC v8; Stage IA Ovarian Cancer AJCC v8; Stage IA Uterine Corpus Cancer AJCC v8; Stage IA1 Cervical Cancer AJCC v8; Stage IA2 Cervical Cancer AJCC v8; Stage IB1 Cervical Cancer AJCC v8; Stage IC Ovarian Cancer AJCC v8
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms | interventions — Delivery of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (focus group, survey): FOCUS GROUP: Patients attend an audiotaped focus group over 90 minutes to provide feedback for survey development.
  SURVEY VALIDATION: Patients complete an online survey over 15-30 minutes at baseline and 2 days later.
  TELEPHONE SURVEY: Patients complete a telephone survey.
  Interventions: Behavioral: Healthcare Activity; Other: Survey Administration

INTERVENTIONS:
Behavioral: Healthcare Activity — Attend focus group
  Other Names: Health Care Activity; Healthcare
Other: Survey Administration — Complete survey

SUMMARY:
This study develops infertility survey among reproductive age women with gynecological and breast cancer. This study aims to learn how women consider whether or not to try to have a baby after surviving cancer. The advice gathered from this survey may be shared with patients and survivors in the future, so that they have information to inform their decisions about cancer treatment and family planning.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To tailor the National Fertility Barriers (NFB) Survey for women who have had gynecological and breast cancers.

II. To administer the tailored survey and evaluate if utilization of infertility clinics and treatments is associated with pregnancies leading to live births after gynecological or breast cancer.

SECONDARY OBJECTIVE:

I. To evaluate whether potential covariates are associated with utilization of infertility clinics and live births after gynecological and breast cancers (e.g. socio-demographic, clinical, psychological, lifestyle, and decision-making characteristics).

OUTLINE:

FOCUS GROUP: Patients attend an audiotaped focus group over 90 minutes to provide feedback for survey development.

SURVEY VALIDATION: Patients complete an online survey over 15-30 minutes at baseline and 2 days later.

TELEPHONE SURVEY: Patients complete a telephone survey.

ELIGIBILITY:
Inclusion Criteria:

* FOCUS GROUP: Women seen at the MD Anderson Oncofertility Clinic and Adolescent and Young Adult Program who are 18-45 years old at the time of cancer diagnosis
* SURVEY VALIDATION: Women seen at the MD Anderson Oncofertility Clinic and Adolescent and Young Adult Program who are 18-45 years old at the time of cancer diagnosis
* TELEPHONE SURVEY: Women in the California Cancer Registry
* TELEPHONE SURVEY: Are 18-45 years old
* TELEPHONE SURVEY: Were diagnosed with early-stage ovarian (IA and IC), endometrial (IA), cervical (IA1-IB1), or breast cancer (I-III)
* TELEPHONE SURVEY: Are 5-12 years post diagnosis between the years of 2007-2014
* TELEPHONE SURVEY: Underwent fertility-preservation treatments

Exclusion Criteria:

* FOCUS GROUP: Do not speak English or Spanish
* SURVEY VALIDATION: Do not read and understand English
* TELEPHONE SURVEY: Do not speak English or Spanish

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women seen at the MD Anderson Oncofertility Clinic and Adolescent and Young Adult Program or women in the California Cancer Registry
Sampling Method: Non-Probability Sample
Enrollment: 1410 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Underlying constructs | Up to 3 years
  Will be measured by the Oncofertility Barriers Scale. Will perform factor analysis using principal axis factoring with oblique rotation to simplify the construct interpretation.
Known-group validity | Up to 3 years
  Will use t-test to compare two groups. If the distributional assumptions are not met, will use the Mann Whitney test.
Convergent validity | Up to 3 years
  Will correlate Oncofertility Barriers Scale scores with Evaluation and Nurturing Relationship Issues, Communication and Happiness scores. Analysis of variance will be used to generate a generalizability coefficient for relevant factors, as distributions allow. As distributions allow, will also assess a priori hypotheses that divergence will be observed among groups of women with different ages, cancer types, time since completing cancer treatment, and priori fertility concerns, as well as access to and utilization of fertility care. All tests will be two-sided and use a significance level of 0.05.
Live birth | Up to 3 years
  Will compare cancer diagnosis, treatment characteristics and patient reported survey results by live birth (yes versus no) using a 2-sample t-test (or Wilcoxon depending on underlying distribution) and chi-squared test (or Fisher's exact test). Will also conduct logistic regression analysis regressing live birth on predictors of interest, and build a multivariable model based on univariate results including all terms significant at the 0.10 level then refining the model using backwards selection to include variables significant at the 0.05 level in the final model.

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Rauh-Hain, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org